CLINICAL TRIAL: NCT02863029
Title: Defining the Role of the Gut Microbiome in Mediating the Effects of Obesity on Intestinal Stem Cells
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-003158
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Obesity
Keywords: Intestinal stem cells
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flexible Sigmoidoscopy (Other): Participants will undergo an unsedated Flexible Sigmoidoscopy in order to obtain 12 mucosal biopsies. Serum cholesterol, triglyceride and HBA1C levels will be determined. Plasma, serum and whole blood will be stored for future use for next generation sequencing and metabolomics to determine the effect of different genetic loci on composition and function of gut microbiota
  Interventions: Procedure: Flexible Sigmoidoscopy

INTERVENTIONS:
Procedure: Flexible Sigmoidoscopy — A sigmoidoscopy is the minimally invasive medical examination of the large intestine from the rectum through the last part of the colon, using a flexible endoscope.

SUMMARY:
New studies are revealing how a high-fat diet could be making the cells of the intestinal lining more likely to become cancerous. The investigators would like to study how obesity influences growth of intestinal stem cells, which could then trigger intestinal tumors.

The investigators are proposing a Pilot Study of 20 subjects (comprised of 10 participants from each of two different BMI categories: 20-25 and 35 & above), who will be asked to provide blood, stool, & urine samples, undergo a flexible sigmoidoscopy, and complete food frequency questionnaires

DETAILED DESCRIPTION:
Hypothesis:

The investigators will test the hypothesis that the gut microbiome drives many of the effects that a pro-obesity high-fat diet has on intestinal stem cell (ISC) biology, which includes 1) an increase in ISC numbers and proliferation, 2) a reduced dependency on niche cells for intestinal organoid initiation, or 3) the acquisition of organoid-initiation by non-stem cell population in the intestinal epithelium.

Specific Aims:

1. To determine whether differences in the gut microbiome in obese human subjects correlates with enhanced intestinal stem cell numbers and function.
2. To validate whether obesity-driven changes in the gut microbiome of human recapitulate the effects of obesity on intestinal stem cell function in germ-free mice.

ELIGIBILITY:
Subject and Control Inclusion Criteria

1. Participants have a Body Mass Index (BMI) between 20-25 or 35 and above.
2. Adults aged 18-65

Exclusion Criteria:

1. Known diagnosis of inflammatory bowel disease, microscopic colitis, celiac disease or other inflammatory conditions or diabetes mellitus
2. Antibiotic use within the past 4 weeks (they can be enrolled after a four week washout period and subsequent use during the 6 month study duration does not exclude them)
3. Bowel preparation for colonoscopy within the past week
4. Significant bowel surgery other than hysterectomy or appendectomy
5. Pregnancy or plans to become pregnant within the study time frame
6. Any other disease(s), condition(s) or habit(s) that would interfere with completion of study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes.
7. Age<18 or vulnerable adults -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Changes in the growth of intestinal stem cells | Two years
  The gut microbiome is altered in obesity and studying intestinal stem cells will be helpful in learning what triggers intestinal tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Purna C Kashyap, M., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Tissue samples will be sent to the Massachusetts Institute of Technology (MIT)

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials